CLINICAL TRIAL: NCT02277275
Title: Effects of a BCAA-supplemented Hypocaloric Diet Versus a Standard Hypocaloric Diet on Weight Loss, Lean Mass Preservation and Improvement of Insulin Sensitivityand Its Benefits Over a High-protein Hypo-caloric Diet.
Brief Title: Comparison of Different Weight Loss Diets With Different Protein Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Lee Yung Seng, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CIRG041
Record Dates: First submitted 2014-10-19; First posted 2014-10-28 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Weight Loss; Insulin Resistance
Keywords: Branched chain amino acid, high protein diet, weight loss
MeSH Terms: conditions — Weight Loss; Insulin Resistance | interventions — Starch

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard protein diet with placebo (Placebo Comparator): Subjects will be provided with standard protein diet for four months and corn starch pills(Placebo) for 6 months
  Interventions: Dietary Supplement: Placebo
- Standard protein diet with BCAA (Experimental): Branched chain amino acid(BCAA) pills will be provided to subjects 0.15g/kg of body weight per day for six months, standard protein diet will be provided for four months
  Interventions: Dietary Supplement: BCAA
- High protein diet with placebo (Placebo Comparator): Subjects will be provided with high protein diet for four months and corn starch pills(Placebo) for 6 months
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BCAA — Branched chain amino acid(BCAA) pills will be provided to subjects 0.15g/kg of body weight per day for six months
  Other Names: AST BCAA 4500
  Arms: Standard protein diet with BCAA
Dietary Supplement: Placebo — Placebo will be provided to the other two arms for six months
  Other Names: Starch pill manufactured to mimic AST BCAA 4500
  Arms: High protein diet with placebo; Standard protein diet with placebo

SUMMARY:
High-protein diets better preserve lean mass than conventional low-fat diets. However, they are costly and have potential health risks. Preserving lean mass is important for sustaining high resting energy expenditure, leading to greater initial weight loss, better weight maintenance and improving blood sugar levels. Branched-chain amino acids (BCAA) supplements are known to preserve lean mass but their effects during weight loss have not been examined. Investigators want to investigate if a BCAA-supplemented diet is more effective than a standard hypocaloric diet in terms of the aforementioned benefits, and yet has less detrimental effects than a high-protein diet for weight loss. Using a 16-week weight loss and 8-week weight maintenance intervention, overweight and obese men and women will be randomized to either a hypocaloric diet with BCAA or placebo supplements or a high-protein diet with placebo supplements. Participants' compliance to the diet versus supplements will be compared. Body composition, resting and diet-induced energy expenditure, insulin sensitivity will be measured and blood samples taken before and after weight loss. These findings will inform on the benefits of BCAA-supplementation during energy restriction and may offer an alternative cost-effective strategy for weight loss and maintenance, without the adverse health effects of a high-protein load.

DETAILED DESCRIPTION:
The prevalence of obesity globally and in Singapore continues to rise despite increased public awareness and efforts to control weight. Its association with chronic metabolic diseases, including diabetes, hypertension, cardiovascular diseases, signify the serious implications of obesity on public health. There remains, however, no scientific consensus on the optimal methods for weight loss and its maintenance over longer periods of time. The Atkins diet was introduced in the late 1990s and has since fuelled the popularity of using high-protein diets for weight loss. Scientific evidence have since shown high-protein diets to be more effective than conventional low-fat, high-carbohydrate diets in producing greater weight loss, at least in the short-term. More importantly, high-protein diets also reduce the amount of lean tissue lost during weight loss and may help to maintain weight loss to a greater extent than conventional diets. However, high-protein diets are also known to raise esterol, albeit improving TG and HDL-cholesterol levels. This could be due to the higher amounts of saturated fats that accompany foods rich in animal protein. In addition, high-protein diets may lower bone mineral density and impact on kidney function. High-protein diets are also more expensive than conventional low-fat, high carbohydrate foods , which is an important consideration for longer term compliance.

Supplements containing branched-chain amino acids (BCAA:leucine, isoleucine and valine) are commonly used among muscle builders and athletic community. BCAAs have been shown to stimulate protein synthesis and preserve lean mass. While a few studies have examined BCAA supplementation with low protein diets for weight loss and found depletion of other essential amino acids, the effects of BCAA supplementation with moderate-protein hypocaloric diets on lean mass preservation during weight loss in energy-restricted obese patients has, to our knowledge, not been investigated. Compared to consuming a high (animal) protein diet, which is also rich in BCAAs, taking BCAA supplements would be a much more convenient and affordable way to obtain similar if not greater quantities of BCAA, without the adverse health effects of a high-protein load on the body.

In this study investigators primarily aim to investigate in overweight/obese subjects, whether a BCAA-supplemented (moderate-protein) hypocaloric diet (BCAA) when compared to a standard (moderate-protein) hypocaloric diet (CT) will result in greater lean mass preservation, resting and diet-induced energy expenditure, and improved insulin sensitivity. Investigators will also examine the effects on lean mass preservation and insulin sensitivity changes between BCAA-supplemented diet and high-protein hypocaloric diet (HP). As a secondary aim, investigators have also powered the study to examine if the BCAA-supplemented diet has added advantage to the high-protein diet by incurring less negative effects on bone mineral density and renal function.

In addition, investigators will determine the participant's compliance to the diet versus supplements as a weight loss and maintenance strategy. The findings of this study will provide us novel insight on BCAA-supplementation in the hypocaloric diet. If this study is successful, BCAA-supplementation on a hypocaloric diet could provide an alternative to a standard (moderate-protein) hypocaloric diet for weight reduction strategy without the attending potential health risks of a high protein load e.g. reduced bone mineral density and detrimental effects on renal function.

There are three main hypotheses which investigators propose to examine.

Hypothesis 1: A BCAA-supplemented hypocaloric diet (BCAA) would lead to greater lean mass preservation during weight loss compared to a standard (moderate-protein) hypocaloric diet (CT).

Diets with varying diet composition, including low-fat, high-carbohydrate diets to high-protein, low-carbohydrate diets have been tested in search of the optimal macronutrient composition for weight loss. High-protein diets have been highly favored for their ability to initiate greater initial weight loss. However, accumulative data from recent studies has shown no significant differences in amount of weight loss between high-protein diets and other traditional (normally low-fat, high-carbohydrate) energy-restricted diets in the longer term (16 weeks to 1 year). It appears that total energy intake, rather than diet composition, is the most important determinant of longer term weight loss.

However, an overriding advantage of high-protein diets is their favorable effects on body composition, that is preserving greater lean mass, compared to high-carbohydrate diets, during weight loss in adult obese patients, independent of energy intake. A recent meta-analysis demonstrated that high protein diets (protein > 1.05g/kg body weight) are associated with up to 1.21 kg additional fat-free mass retention compared with diets of lower protein intake. Lean mass or fat-free mass is a main determinant of basal (resting) energy expenditure. Its greater preservation would reduce the weight loss-induced decreased in energy expenditure, which might have two important implications. Firstly, higher basal energy expenditure during weight loss could lead to greater weight loss for the same amount of calories consumed. Secondly, the amount of lean mass preserved at the end of weight loss might mitigate weight regain during maintenance phase of weight loss, i.e. success of weight maintenance.

Branched-chain amino acids like leucine, isoleucine and valine are substrates for protein synthesis and also potent nutrients that regulate protein metabolism. Supplementation with leucine or leucine-rich protein sources have been suggested to develop muscle mass or prevent protein loss in conditions characterized by muscle protein wasting. In human studies, the use of leucine or leucine-rich protein sources supplementation have been well-investigated to optimize the effects of exercise on body composition.Several studies have examined the impact of chronic (average of 3 months) leucine-rich amino acid supplementation in healthy elderly humans, and have demonstrated significant improvement in lean body mass, muscle strength and physical capacity.

Whether the lean mass preservation during high-protein hypocaloric diet is due to the presence of the higher amounts of BCAA content is less clear. Two studies have examined the use of whey protein (rich in BCAA) in weight loss but it was uncertain if the benefits of enhanced weight loss with less lean muscle loss can be attributed to the BCAA alone or due to the enrichment of other nutrients like calcium and bioactive peptides in the whey protein fraction. It is also not clear whether animal sources of protein (rich in BCAAs) are more beneficial than plant sources of protein on energy expenditure, body composition , satiety and fat loss.

To investigators' knowledge, no studies have specifically examined the beneficial effect of BCAA supplementation with a moderate-protein diet on lean mass preservation during weight loss in energy-restricted obese patients. Investigators hypothesize that similar to a high-protein diet (as shown in literature), a BCAA-supplemented hypocaloric diet would also lead to greater lean mass preservation than a standard (moderate-protein) hypocaloric diet during weight loss. In addition, investigators want to examine the effects on lean mass preservation between BCAA-supplemented hypocaloric diet and high protein hypocaloric diet.

Hypothesis 2: Improvement in insulin sensitivity with a BCAA-supplemented hypocaloric diet (BCAA) is greater than a standard (moderate-protein) hypocaloric diet (CT).

The insulin stimulating effects of proteins maybe mediated through specific amino acids, making them potent modulators of insulin action and glucose metabolism. In animal models, BCAA supplementation has been found to improve glucose tolerance and stimulate glucose uptake in skeletal muscle by mechanisms involving glycogen synthase activity. While energy restriction and weight loss have positive effects on insulin sensitivity , whether diet composition further impacts on insulin sensitivity is still inconclusive. Several studies found significant improvement in insulin sensitivity after high-protein diets compared to control diets, independent of weight loss, while others did not. As skeletal muscle mass is a major determinate of insulin sensitivity, investigators postulate that due to greater lean mass preservation, the BCAA diet would result in greater improvement in insulin sensitivity compared to CT diet.

Hypothesis 3: The BCAA-supplementation diet (BCAA) would be easier to adhere to and has less detrimental effects on bone mineral density and renal function than the high-protein diet (HP), leading to better (short-term) weight maintenance and less weight regain.

Maintaining weight loss is a greater challenge than the weight loss process and may not be as easily achieved. Studies have shown that weight regain is significantly lesser in subjects in the high-protein group compared to control group after six months to a year on a weight-maintenance diet. In these studies, study foods are provided and may not reflect real-life free-living situations during weight maintenance phase. Achieving a high-protein diet long term can be costly and requires careful planning of meals. To what extent subjects can continue to maintain the same diet composition as their weight loss diet on their own accord at energy balance during weight maintenance has not been well-investigated The effectiveness of longer term BCAA supplementation in hypocaloric diet has also not been fully investigated. If BCAA supplementation could induce similar metabolic improvement as of a high-protein diet during the weight loss phase, it might help to maintain body weight through easy administration and greater compliance in the longer term.

In this study, investigators proposed to provide BCAA supplements to the BCAA group and placebo supplements provided to the HP and CT groups throughout the entire study (weight loss and maintenance phases).

Study foods will, however, only be provided during the weight loss phase. Investigators speculate that overall, adherence to supplementation would be better than adherence to the respective diet compositions at the end of the weight maintenance phase for subjects in all three groups. Investigators hypothesize that while subjects on the HP and BCAA diets will have less weight regain in the initial weight maintenance phase (due to greater lean mass) than the CT group, the BCAA group will have the least weight regain at the end of weight maintenance phase due to better compliance.

Concerns have been raised over the safety of high-protein diets. Studies have indicated that increase protein intake is associated with increased renal calcium excretion, negative calcium balance, bone resorption and causes hyperfiltration. At the same time, it is also known that loss of bone mass often accompanies weight loss induced by calorie restriction. Whether high-protein diets have a detrimental impact on bone mineral density and renal function is still inconclusive. In this study, investigators hypothesize that the BCAA-supplemented diet would result in lesser detrimental effects on bone mineral density and renal function than the high-protein diet.

Other secondary hypotheses:

The three dietary interventions may lead to significant differences in markers of cardiometabolic outcomes including inflammatory markers

The resting/basal metabolic rate change with time, and diet induced thermogenesis, may differ between the three groups

The resting basal metabolic rate change in the subjects with weight loss at 16 weeks predicts the weight gain/rebound at 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to comply with study procedures and given written informed consent
2. Chinese, aged 21-45 years old
3. Body mass index (BMI) between 25 -35 kg/m2 and % body fat of more than 25 %.
4. Sedentary adults, with <1 episode of exercise per week
5. Not have a history of food allergies or food intolerances
6. Have maintained a stable body weight for at least 3 months prior to the study.
7. Be a non-smoker
8. Drinks less than 3 caffeinated beverages per day (coffee/tea/energy drinks)
9. Drinks less than 3 units of alcohol per day

Exclusion Criteria:

1. Subjects with diabetes, renal impairment, high blood pressure, gastrointestinal problems, asthma, eczema, anaemia or on medications that will affect glucose metabolism (e.g. corticosteroids) or lipid metabolism/insulin resistance (e.g. niacin, fibrates, metformin) and other significant medical conditions, which in the investigator's opinion would confound interpretation of results.
2. Recent changes (gain or loss) in weight of >5% over the past 3 months
3. Significant changes in diet over the past 3 months
4. Any use of weight-reduction drugs in the past 6 months
5. Use of any prescription medication that cannot be safely discontinued within 14 days prior to study entry
6. Have special dietary needs/restrictions e.g. vegetarian diet or unable to consume fish, seafood and beef
7. History of eating disorders or irregular eating habits
8. High level of physical activity (exercise > 5hr per week)
9. Women who are pregnant and lactating and women of reproductive age group who plan to conceive within 6 months. A pregnancy test will be performed for women in the reproductive age group.
10. Have contraindications to Magnetic Resonance Imaging (MRI) that includes metallic implants, pacemakers or stimulators, or any other methodology applied in the study.
11. Have been involved in any clinical or food study within the preceding month.
12. Presently consuming amino acid or protein-related supplements.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Changes in body compostion(i.e muscle mass, fat mass) by DEXA scan measurements | Week 0, 16 and 24
  lean mass, fat mass

SECONDARY OUTCOMES:
Changes in resting and diet-induced energy expenditure | Week 0, 16 and 24
  Energy expenditure will be measured using indirect calorimetry before and after consuming the test meal
Changes in insulin resistance | Week 0, 16 and 24
  Insulin sensitivity index can be derived from HOMA-IR and Masuda method
inflammatory markers and gene expressions of PBMC | week 0, 16, 24

CONTACTS AND LOCATIONS:
Overall Officials: Yung Seng Lee, Principal Investigator — Associate Professor
Locations (1):
- Clinical Nutrition Research Center, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No